CLINICAL TRIAL: NCT06569446
Title: Understanding the Barriers to Rectal Irrigation in Patients With Defaecatory Dysfunction
Brief Title: Barriers to Rectal Irrigation in Defaecatory Dysfunction
Status: Not yet recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 336619
Record Dates: First submitted 2024-08-21; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-02

CONDITIONS: Defecation Disorder; Constipation - Functional; Constipation by Outlet Obstruction; Faecal Incontinence; Faecal Smearing; Obstructive Defecation Syndrome
Keywords: chronic constipation; rectal irrigation; trans-anal irrigation; evacuation disorders; faecal incontinence; barriers; patient interviews; structured interviews
MeSH Terms: conditions — Encopresis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Focused Group Sessions: This will involve semi-structured, open-ended questions about hypothesized barriers to rectal irrigation where the interviewer will ask a pre-determined number of questions and the participants will answer which will further initiate discussion allowing new themes to emerge. After the entire list of barriers is discussed, participants will be asked if they have any new barriers to add which have not been discussed. All new barriers identified will be added to the hypothesized barriers list for the next focused group sessions. Focused group sessions will continue until no new barriers are found in two consecutive sessions (thematic saturation).
  Interventions: Other: There is no intervention. This a qualitative study to explore barriers to rectal irrigation
- Cognitive Interviews: This will involve semi-structured, open-ended questions about barriers to rectal irrigation identified during focused group sessions where the interviewer will ask pre-determined number of questions for individual participants to answer.
  Interventions: Other: There is no intervention. This a qualitative study to explore barriers to rectal irrigation

INTERVENTIONS:
Other: There is no intervention. This a qualitative study to explore barriers to rectal irrigation — This will involve semi-structured, open-ended questions about hypothesized barriers to rectal irrigation where the interviewer will ask a pre-determined number of questions and the participants will answer which will further initiate discussion allowing new themes to emerge. After the entire list of barriers is discussed, participants will be asked if they have any new barriers to add which have not been discussed. All new barriers identified will be added to the hypothesized barriers list for the next focused group sessions. Focused group sessions will continue until no new barriers are found in two consecutive sessions (thematic saturation).
  9.2 Phase - 2 includes Cognitive Interviews This will involve semi-structured, open-ended questions about barriers to rectal irrigation identified during focused group sessions where the interviewer will ask pre-determined number of questions for individual participants to answer.

SUMMARY:
Rectal irrigation is the introduction of warm tap water through the anal canal into the rectum to initiate defaecation. NICE recommends that rectal irrigation be considered in patients with constipation(1) and faecal incontinence (2) refractory to conservative measures such as lifestyle advice and pharmacological therapy, and bio-feedback therapy which is a treatment to help patients learn to strengthen or relax their pelvic floor muscles to improve bowel or bladder function by retraining the pelvic floor muscles and provides psychosocial support(3). Studies have shown that up to half patients discontinue rectal irrigation within a year of commencing therapy (4) (5). The investigators want to understand barriers to rectal irrigation by conducting focused group sessions and cognitive interviews of patients who have used or declined rectal irrigation.

DETAILED DESCRIPTION:
Rectal irrigation is the introduction of warm tap water through the anal canal into the rectum to initiate defaecation. Proposed mechanisms of action include simple mechanical washout, colonic movement stimulated by the washout, or a combination of these(1).

By regularly emptying the bowel in this manner, rectal irrigation helps re-establish control of bowel function and enables the patients to choose the time and place of evacuation thus re-instating more predictable bowel movement (2) and therefore allowing them to have a better quality of life.

National Institute for Health and Care Excellence recommends that rectal irrigation be considered in patients with constipation(8) and faecal incontinence (9) refractory to conservative measures such as lifestyle advice and pharmacological therapy, and bio-feedback therapy which is a treatment to help patients learn to strengthen or relax their pelvic floor muscles to improve bowel or bladder function by retraining the pelvic floor muscles and provides psychosocial support(10).

Studies have looked at outcomes of rectal irrigation in patients with defaecatory difficulties (6,11,12) where improvement in symptoms or quality of life in patients after using irrigation has been reported. Christensen reported that 52% of the patients used rectal irrigation for a median of 8 months before discontinuing treatment(11) where reasons for discontinuation were unsatisfactory effect, faecal incontinence, time consumption, disliking for treatment, side effects, leakage of irrigation fluid and expulsion of rectal catheter. Tamvakeras reported four (22%) out of eighteen patients discontinued rectal irrigation in a median length of 4.8 months. Three of the four patients who discontinued rectal irrigation found it ineffective while the fourth patient discontinued due to resolution of symptoms(12).

Barriers to using rectal irrigation other than side-effects or unsatisfactory outcome still need to be explored such as cultural or social reasons and lack of knowledge or fear about the treatment.

The investigators aim to organize focused group sessions and cognitive interviews of patients to understand the barriers to irrigation so that these can be addressed for better compliance and outcome leading to a better quality of life in patients with defaecatory difficulties.

9. Study design This is a qualitative study which has two phases.

11.2 Participant Recruitment After screening, research will be introduced to the eligible participants by a member of the clinical team during their bowel function clinic appointment (face-to-face / telephone). Participant information sheet will be provided or posted depending on type of appointment. Patient details will be noted on eligibility log and passed on to the research team. It will be ensured that the investigators have a fair selection of patients by stratifying them based on gender, age, ethnicity, socio-economic status and presenting complain. This will be to make sure our research cohort is as close to the actual population as possible. For e.g., the investigators will ensure that there is equal representation of all types of ethnicity and socio-economic groups. Patients will be given at least 48 hours to consider participation and will be contacted over the phone by a member of the research team. Should patients require more time to think, then another call will be arranged as per their convenient time. The call will be to discuss the research and answer any queries the patients may have following which, if the patients are happy to participate they will be invited to the focused group sessions or cognitive interviews depending on what phase of the study they are being recruited for. Should they decide not to participate, they will be reassured that it will not have any impact on their on-going care in the department. A hospital interpreter will be arranged for patients with limited English communication skills to help with consenting, attending focused group sessions and cognitive interviews. For group sessions, if an interpreter is required, all participants will be notified via a telephone call before the session and consent will be obtained and documented.

For those unable to read or write, a witness from the participant's family or a carer can be arranged to come into the face-to-face appointment with the participant, however consent will have to be provided by the participant. Patients attending face-to-face group will be consented before starting the session on the day by a member of the research team while those attending online focused group sessions will be sent e-consent forms via encrypted NHS email by a member of the research team. E-consent forms will be required to be returned via email.

11.3 Schedule of appointments

Focused Group Session - Phase 1 of study Two types of focused groups will be co-ordinated according to participant's convenience and availability. Group 1 will include participants who are currently using rectal irrigation or have used in the past. Group 2 will include participants who had declined rectal irrigation. Four participants will be recruited for each of the two groups. Since the pelvic floor unit receive referrals from both urban and rural communities, it may not be feasible for all participants to travel for the group sessions, or some participants may feel embarrassed to attend and participate in discussion with others or feel nervous about travelling due to symptoms such as faecal incontinence. Therefore, to facilitate, the investigators will organise both in person and virtual focused group sessions if need be. Face to face group sessions will be conducted in Pelvic Floor Unit at St. Thomas' Hospital while virtual sessions will be conducted on Microsoft Teams. Participants wanting to attend virtually will be asked for their email address to send the invitation and consent to.

Each focused group will be facilitated by a member of the research team. This session will last up to 60 minutes. Following introductions, a list of hypothesized barriers (HB) to using rectal irrigation will be distributed and each item on the list will be discussed by facilitator first asking a pre-determined question. HB will include reasons identified by previous studies for discontinuing rectal irrigation(11,12) along with factors the investigators think may contribute as barriers. With discussions in the focused group sessions, the investigators hope to discover more barriers to rectal irrigation from participants which will be added to the list for next focused group session. At the end, all participants will be asked if they are aware of any barriers which have not been covered in the session and these will be noted. After the session, a twenty-minute talk to educate patients on rectal irrigation will be offered, should participants wish to attend. Focused group sessions will continue until a barrier saturation (no more new barriers found upon discussion in two consecutive focused group sessions) is reached. Male and female participants will be assigned to separate interview groups to avoid embarrassment should the participants feel that way and find it difficult to have an open discussion.

Virtual sessions will be conducted via Microsoft teams which will be both audio and video recorded. Participants can turn off their cameras if they do not wish to be visually recorded. This will be reminded at the start of the virtual session. All face-to face focused group sessions will be audio recorded via trust encrypted recording device and transcribed. At the end of the session, the recording from both audio encrypted recording device and recording from Microsoft teams will be listened to and transcribed by the facilitator. Participants quotes will be pseudonymised such that each participant will be assigned a registration number upon recruitment by a member of the research team for e.g. BRI-001. Once the summary is prepared from the transcribed notes then the audio recording and Microsoft Teams recording will be destroyed as per the sponsor's instructions. Until the investigators destroy them , the data will be stored in the Trust computer and devices in locked cabinets in accordance with Data Protection act 2018 and the NHS Confidentiality Code of Practice.

Cognitive Interviews - Phase 2 of study Ten individuals who have not participated in phase 1 of the study will be invited to attend cognitive interviews. This will be to validate the barriers discovered during focused group sessions. These sessions be conducted as described in line with the process described in phase 1 for the focus groups, with the option of face-to-face or virtual sessions. However unlike with the focus groups, these will be one to one sessions .

Strength This is the first study to identify and understand barriers to rectal irrigation via qualitative interviews other than complications of using the irrigation device and no improvement in symptoms. It is a patient centred study to help inform clinicians about barriers to rectal irrigation faced by patients. This can help take measures in future for resolution of barriers to have better outcomes and patient compliance to treatment. Focused group sessions followed by educational session will also help create more awareness amongst our patients regarding using rectal irrigation. It will also allow patients to feel more involved in their care and their problems regarding the treatment being listened to.

Data

12.1 Data to be collected

Personal data Identifiable patient data will be recorded only for the purpose of contacting patients for e.g., name, date of birth and address, and will be kept confidential in a password protected file (Microsoft Excel) by the principle investigator (PI) and co-investigator (TG) where no third party will have access to it.

Socio-demographics The co-investigator (TG) will assign a research registration number to each participant after recruitment and consenting such as BRI-001. All socio-demographic data will be collected against this registration number to pseudonymise data for analysis. Socio-demographic data will include age, gender, post code to calculate proxy marker for socio-economic status and commute distance, ethnicity and mode of transport to the hospital if coming for face-to-face session/interview.

Transcribed data All representative quotes recorded and transcribed will be pseudonymised with any identifiers revealed being replaced with the participants registration number such as BRI-001.

13 End of the study definition The study will be considered to have come to an end when the last patient (tenth) of Phase-2 of the study has undergone cognitive interview.

ELIGIBILITY:
Inclusion Criteria:

* Patients who

  1. are/have

     1. currently using rectal irrigation
     2. have previously used rectal irrigation
     3. declined rectal irrigation
  2. equal to or over 18 years
  3. have defaecatory difficulties
  4. Failed nurse-led biofeedback treatment
  5. have ability and willingness to give informed consent

     Exclusion Criteria:

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The following patients will be excluded:
  * Lack capacity
  * Unable to participate in discussion
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Barriers to rectal irrigation | 60 minutes
  To understand the barriers to rectal irrigation in patients with defaecatory dysfunction by conducting focused group sessions.

SECONDARY OUTCOMES:
Validate barriers to rectal irrigation | 60 minutes
  To validate the barriers discovered during focused group sessions by conducting cognitive interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Hainsowrth, FRCS, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Christensen P, Krogh K. Transanal irrigation for disordered defecation: a systematic review. Scand J Gastroenterol. 2010 May;45(5):517-27. doi: 10.3109/00365520903583855. PMID 20199336
- [Background] Krogh K, Ostergaard K, Sabroe S, Laurberg S. Clinical aspects of bowel symptoms in Parkinson's disease. Acta Neurol Scand. 2008 Jan;117(1):60-4. doi: 10.1111/j.1600-0404.2007.00900.x. PMID 18095955
- [Background] Shandling B, Gilmour RF. The enema continence catheter in spina bifida: successful bowel management. J Pediatr Surg. 1987 Mar;22(3):271-3. doi: 10.1016/s0022-3468(87)80345-7. PMID 3550032
- [Background] Briel JW, Schouten WR, Vlot EA, Smits S, van Kessel I. Clinical value of colonic irrigation in patients with continence disturbances. Dis Colon Rectum. 1997 Jul;40(7):802-5. doi: 10.1007/BF02055436. PMID 9221856
- [Background] Gardiner A, Marshall J, Duthie G. Rectal irrigation for relief of functional bowel disorders. Nurs Stand. 2004 Nov 10-16;19(9):39-42. doi: 10.7748/ns2004.11.19.9.39.c3755. PMID 15574053
- [Background] Crawshaw AP, Pigott L, Potter MA, Bartolo DC. A retrospective evaluation of rectal irrigation in the treatment of disorders of faecal continence. Colorectal Dis. 2004 May;6(3):185-90. doi: 10.1111/j.1463-1318.2004.00584.x. PMID 15109384
- [Background] Pakzad M, Telford K, Ward K, Keighley M. Seizing the opportunity to improve patient care: pelvic floor services in 2021 and beyond. Br J Hosp Med (Lond). 2021 Sep 2;82(9):1-3. doi: 10.12968/hmed.2021.0387. Epub 2021 Sep 16. PMID 34601937
- [Background] Christensen P, Krogh K, Buntzen S, Payandeh F, Laurberg S. Long-term outcome and safety of transanal irrigation for constipation and fecal incontinence. Dis Colon Rectum. 2009 Feb;52(2):286-92. doi: 10.1007/DCR.0b013e3181979341. PMID 19279425
- [Background] Tamvakeras P, Horrobin C, Chang J, Chapman M. Long-Term Outcomes of Transanal Irrigation for Bowel Dysfunction. Cureus. 2023 Jul 26;15(7):e42507. doi: 10.7759/cureus.42507. eCollection 2023 Jul. PMID 37502470
- See also: NICE guidelines for management of faecal incontinence in adults — https://www.nice.org.uk/guidance/cg49/chapter/Recommendations
- See also: Biofeedabck — http://www.pelvicfloorcenter.org/content/biofeedback